CLINICAL TRIAL: NCT00827619
Title: Evaluation of the Zilver® Flex™ Vascular Stent in the Above-the-Knee Femoropopliteal Artery
Brief Title: Zilver® Flex™ Vascular Stent Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-009; 100005, ZBLL
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Peripheral Arterial Disease (PAD)
Keywords: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Stents; Mutagenesis, Insertional

ARMS (1):
- 1 (Other): single arm non-randomized post-market study
  Interventions: Device: Zilver® Flex™ Vascular Stent

INTERVENTIONS:
Device: Zilver® Flex™ Vascular Stent — Stenting of the Above-the-Knee Femoropopliteal Artery
  Other Names: Stenting; Vascular Stent; Implant

SUMMARY:
This study is intended to evaluate the long-term effectiveness of treatment of de novo or restenotic lesions of the above-the-knee femoropopliteal artery using the Zilver® Flex™ Vascular Stent which has received the CE mark for commercial use. The study is designed as a single arm non-randomized post-approval study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years old and have at least 1 stenotic atherosclerotic lesion of the above-the-knee femoropopliteal artery may be considered for enrollment.
* To be enrolled in the study, the lesion must be the appropriate size and and no prior stent in the target vessel may be present.

Exclusion Criteria:

* Patient is < 18 years of age.
* Patient is pregnant or breast-feeding.
* Patient is simultaneously participating in an investigational drug or device study. The patient must have completed the follow-up phase for the primary endpoint of any previous study at least 30 days prior to enrollment in this study.
* Patient has had previous stenting of the target vessel.
* Patient has a medical condition or disorder that would limit life expectancy to less than 1 year or that may cause noncompliance with the protocol or confound the data analysis.
* Patient in whom antiplatelet and/or anticoagulant therapy is contraindicated.
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Patient has known hypersensitivity or contraindication to aspirin, antiplatelet medication, contrast dye, or nitinol that, in the opinion of the investigator, cannot be adequately premedicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-02; Primary Completion 2011-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Primary patency of the treated lesion within the superficial femoral artery | 1 year after patient enrollment

SECONDARY OUTCOMES:
Procedural success and primary-assisted and secondary patency, thrombosis/total occlusion rate, clinical improvement, and functional status improvement | 1 year after patient enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ricke, MD, Principal Investigator — Universitatsklinikum Magdeburg
Locations (3):
- Germany (3):
  - Herz-Zentrum, Bad Krozingen
  - Gemeinschaftspraxis, Leipzig
  - Universitatsklinikum Magdeburg, Magdeburg